CLINICAL TRIAL: NCT05016141
Title: Health in Motion- A Digital Fall Prevention Program Designed to be Delivered in the Home
Brief Title: Health in Motion- A Pragmatic Clinical Trial- Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blue Marble Rehab Inc (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AG043191; 2R44AG043191-04A1 (NIH)
Record Dates: First submitted 2021-07-19; First posted 2021-08-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: fall; fall prevention; fall injury; fear of falling; fall efficacy

STUDY DESIGN:
Intervention Model Description: comparative prospective longitudinal (12-months) observational cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no intervention (No Intervention): Participants will be observed for 12 months. Participants will use the Health in Motion app to set goals and keep track of their health and health events, including falls. These participants will NOT receive the education modules or the exercise program.
- digital fall prevention program (Experimental): Participants will complete the Health in Motion digital fall prevention program for 12 months. This program consists of education modules (modified from the Matter of Balance Program) and exercises based on a digital translation of the Otago Exercise Program.
  Interventions: Behavioral: digital fall prevention program

INTERVENTIONS:
Behavioral: digital fall prevention program — The participants will receive a digital fall prevention program consisting of fall risk reduction education (modified Matter of Balance), Otago Exercise Program, Personalized S.M.A.R.T Goals, and will use the app to keep track of their health and health events, including falls.
  Arms: digital fall prevention program

SUMMARY:
Falls among older adults are a serious public health concern and injuries resulting from falls can cause significant loss of independence, premature death, and higher caregiver burden. Home-based fall prevention programs, such as the Otago Exercise Program, educate older adults about the importance of identifying fall risk and provide strategies for reducing fall risk; however, many are costly and are not scalable, accessible, or sustainable. This project will evaluate the use of a digital solution that translates evidence-based fall prevention programs (such as Otago Exercise Program and Matter of Balance) to a digital solution (Health in Motion Fall Prevention Platform), as an alternative to home-based fall prevention programs that is affordable, scales to the millions of older adults across the country at risk for falls and is sustainable for the older adult's life.

DETAILED DESCRIPTION:
This study will involve 2 groups. Both groups will be followed for 12 months. The investigators will use a comparative prospective longitudinal (12-months) observational cohort study to compare the Health in Motion Fall Prevention Program with a no-intervention group. Metrics of effectiveness include the rate of falls, fall risk, fear of falling, and falls efficacy. Economic benefit will be measured using the EQ-5D-5L, along with hospital and clinical visits. The primary outcome is the incidence of falls (rate in person-months).

ELIGIBILITY:
Inclusion Criteria:

* age of 55 and older
* if history of 2 or more falls in the past year with a physician or physical therapist approval
* Score >31 on the TICS (Telephone Interview for Cognitive Screen)
* Easy for Me screen for inclusion

Exclusion Criteria:

* any person who has been told by their physician that they should not exercise

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Rate of Falls per month | Change from baseline fall rate at 3 months
  Number of falls per month / number of participants x 1000
Rate of Falls per month | Change from baseline fall rate at 6 months
  Number of falls per month / number of participants x 1000
Rate of Falls per month | Change from baseline fall rate at 9 months
  Number of falls per month / number of participants x 1000
Rate of Falls per month | Change from baseline fall rate at 12 months
  Number of falls per month / number of participants x 1000

SECONDARY OUTCOMES:
Timed Up and Go Test | Change from baseline at 3 months
  Time taken to stand up from a seated position, walk 10 feet, turn around, return to the chair, sit down
Timed Up and Go Test | Change from baseline at 6 months
  Time taken to stand up from a seated position, walk 10 feet, turn around, return to the chair, sit down
Timed Up and Go Test | Change from baseline at 9 months
  Time taken to stand up from a seated position, walk 10 feet, turn around, return to the chair, sit down
Timed Up and Go Test | Change from baseline at 12 months
  Time taken to stand up from a seated position, walk 10 feet, turn around, return to the chair, sit down
4 Stage Balance Test | Change from baseline at 3 months
  This test measures the ability to stand for 10 seconds in 4 progressively more challenging positions from standing with feet side by side to standing on one leg. The score is equal to the total time taken to achieve the highest level. The maximum score is 40. If a participant is not able to stand with their feet in tandem, they are considered at higher risk of falling.
4 Stage Balance Test | Change from baseline at 6 months
  This test measures the ability to stand for 10 seconds in 4 progressively more challenging positions from standing with feet side by side to standing on one leg. The score is equal to the total time taken to achieve the highest level. The maximum score is 40. If a participant is not able to stand with their feet in tandem, they are considered at higher risk of falling.
4 Stage Balance Test | Change from baseline at 9 months
  This test measures the ability to stand for 10 seconds in 4 progressively more challenging positions from standing with feet side by side to standing on one leg. The score is equal to the total time taken to achieve the highest level. The maximum score is 40. If a participant is not able to stand with their feet in tandem, they are considered at higher risk of falling.
4 Stage Balance Test | Change from baseline at 12 months
  This test measures the ability to stand for 10 seconds in 4 progressively more challenging positions from standing with feet side by side to standing on one leg. The score is equal to the total time taken to achieve the highest level. The maximum score is 40. If a participant is not able to stand with their feet in tandem, they are considered at higher risk of falling.
One Leg Stand Test | Change from baseline at 3 months
  This test measures the ability to stand for on one leg for up to 30 seconds. If a participant is not able to stand for 5 seconds, they are considered at higher risk of falling.
One Leg Stand Test | Change from baseline at 6 months
  This test measures the ability to stand for on one leg for up to 30 seconds. If a participant is not able to stand for 5 seconds, they are considered at higher risk of falling.
One Leg Stand Test | Change from baseline at 9 months
  This test measures the ability to stand for on one leg for up to 30 seconds. If a participant is not able to stand for 5 seconds, they are considered at higher risk of falling.
One Leg Stand Test | Change from baseline at 12 months
  This test measures the ability to stand for on one leg for up to 30 seconds. If a participant is not able to stand for 5 seconds, they are considered at higher risk of falling.
30 Second Sit to Stand Test | Change from baseline at 3 months
  This test measures the number of times a participant can stand up from a seated position in 30 seconds.
30 Second Sit to Stand Test | Change from baseline at 6 months
  This test measures the number of times a participant can stand up from a seated position in 30 seconds.
30 Second Sit to Stand Test | Change from baseline at 9 months
  This test measures the number of times a participant can stand up from a seated position in 30 seconds.
30 Second Sit to Stand Test | Change from baseline at 12 months
  This test measures the number of times a participant can stand up from a seated position in 30 seconds.
Fall Risk Questionnaire | Change from baseline at 3 months
  This is a multi-factorial questionnaire that can be used to predict fall risk. Questions relate to history of falls, gait/balance, muscle weakness, incontinence, sensation/proprioception, depression, vision and medications. The highest (worst) score = 14. A score of 0-3 denotes low fall risk and scores from 4-14 denote higher fall risk.
Fall Risk Questionnaire | Change from baseline at 6 months
  This is a multi-factorial questionnaire that can be used to predict fall risk. Questions relate to history of falls, gait/balance, muscle weakness, incontinence, sensation/proprioception, depression, vision and medications. The highest (worst) score = 14. A score of 0-3 denotes low fall risk and scores from 4-14 denote higher fall risk.
Fall Risk Questionnaire | Change from baseline at 9 months
  This is a multi-factorial questionnaire that can be used to predict fall risk. Questions relate to history of falls, gait/balance, muscle weakness, incontinence, sensation/proprioception, depression, vision and medications. The highest (worst) score = 14. A score of 0-3 denotes low fall risk and scores from 4-14 denote higher fall risk.
Fall Risk Questionnaire | Change from baseline at 12 months
  This is a multi-factorial questionnaire that can be used to predict fall risk. Questions relate to history of falls, gait/balance, muscle weakness, incontinence, sensation/proprioception, depression, vision and medications. The highest (worst) score = 14. A score of 0-3 denotes low fall risk and scores from 4-14 denote higher fall risk.
Activities Specific Balance Confidence Scale 5 Level | Change from baseline at 3 months
  This questionnaire measures the participant's confidence in performing activities of daily living in which each item is rated from 0% (no confidence) to 100% (complete confidence). It correlates with other measures of self-efficacy and balance measures.
Activities Specific Balance Confidence Scale 5 Level | Change from baseline at 6 months
  This questionnaire measures the participant's confidence in performing activities of daily living in which each item is rated from 0% (no confidence) to 100% (complete confidence). It correlates with other measures of self-efficacy and balance measures.
Activities Specific Balance Confidence Scale 5 Level | Change from baseline at 9 months
  This questionnaire measures the participant's confidence in performing activities of daily living in which each item is rated from 0% (no confidence) to 100% (complete confidence). It correlates with other measures of self-efficacy and balance measures.
Activities Specific Balance Confidence Scale 5 Level | Change from baseline at 12 months
  This questionnaire measures the participant's confidence in performing activities of daily living in which each item is rated from 0% (no confidence) to 100% (complete confidence). It correlates with other measures of self-efficacy and balance measures.
VR-12 | Change from baseline at 3 months
  This questionnaire measures quality of life over the past 4 weeks.
VR-12 | Change from baseline at 6 months
  This questionnaire measures quality of life over the past 4 weeks.
VR-12 | Change from baseline at 9 months
  This questionnaire measures quality of life over the past 4 weeks.
VR-12 | Change from baseline at 12 months
  This questionnaire measures quality of life over the past 4 weeks.
European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | Change from baseline at 3 months
  This is a standardized measure of health status for clinical and economic appraisal. The test is a self report health state that domains including mobility, self-care, anxiety/depression, pain/discomfort) using a 5 point scale and a visual analog scale (VAS).
  We will calculate quality-adjusted life years (QALY) using the EQ-5D-5L and the appropriate weights from each instrument to compare differences in the incremental cost-effectiveness ratios.
European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | Change from baseline at 6 months
  This is a standardized measure of health status for clinical and economic appraisal. The test is a self report health state that domains including mobility, self-care, anxiety/depression, pain/discomfort) using a 5 point scale and a visual analog scale (VAS).
  We will calculate quality-adjusted life years (QALY) using the EQ-5D-5L and the appropriate weights from each instrument to compare differences in the incremental cost-effectiveness ratios.
European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | Change from baseline at 9 months
  This is a standardized measure of health status for clinical and economic appraisal. The test is a self report health state that domains including mobility, self-care, anxiety/depression, pain/discomfort) using a 5 point scale and a visual analog scale (VAS).
  We will calculate quality-adjusted life years (QALY) using the EQ-5D-5L and the appropriate weights from each instrument to compare differences in the incremental cost-effectiveness ratios.
European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | Change from baseline at 12 months
  This is a standardized measure of health status for clinical and economic appraisal. The test is a self report health state that domains including mobility, self-care, anxiety/depression, pain/discomfort) using a 5 point scale and a visual analog scale (VAS).
  We will calculate quality-adjusted life years (QALY) using the EQ-5D-5L and the appropriate weights from each instrument to compare differences in the incremental cost-effectiveness ratios.
Education Modules Data (Intervention Group Only) | through study completion, an average of 1 year.
  Time Taken: The Health in Motion App captures data time taken to complete the lessons.
Education Modules Data (Intervention Group Only) | through study completion, an average of 1 year.
  Qualitative Analysis of text entries.
System Usability Scale | Change from baseline at 3 months
  The System Usability Scale is used to evaluate usability and learnability of software products. We will use information from this survey to improve the usability of Health in Motion. The test uses a 0-5 Likert scale. The statements are worded such that the best score alternates between 1 (Strongly Disagree) and 5 (Strongly Agree). For example, statement #1 is "I think that I would like to use this system frequently" whereas statement #2 is "I found this system unnecessarily complex". The participant's scores for each question are converted to a new number, added together, and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  SUS scores above 68 are considered above average and anything below 68 is below average.
System Usability Scale | Change from baseline at 6 months
  The System Usability Scale is used to evaluate usability and learnability of software products. We will use information from this survey to improve the usability of Health in Motion. The test uses a 0-5 Likert scale. The statements are worded such that the best score alternates between 1 (Strongly Disagree) and 5 (Strongly Agree). For example, statement #1 is "I think that I would like to use this system frequently" whereas statement #2 is "I found this system unnecessarily complex". The participant's scores for each question are converted to a new number, added together, and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  SUS scores above 68 are considered above average and anything below 68 is below average.
System Usability Scale | Change from baseline at 9 months
  The System Usability Scale is used to evaluate usability and learnability of software products. We will use information from this survey to improve the usability of Health in Motion. The test uses a 0-5 Likert scale. The statements are worded such that the best score alternates between 1 (Strongly Disagree) and 5 (Strongly Agree). For example, statement #1 is "I think that I would like to use this system frequently" whereas statement #2 is "I found this system unnecessarily complex". The participant's scores for each question are converted to a new number, added together, and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  SUS scores above 68 are considered above average and anything below 68 is below average.
System Usability Scale | Change from baseline at 12 months
  The System Usability Scale is used to evaluate usability and learnability of software products. We will use information from this survey to improve the usability of Health in Motion. The test uses a 0-5 Likert scale. The statements are worded such that the best score alternates between 1 (Strongly Disagree) and 5 (Strongly Agree). For example, statement #1 is "I think that I would like to use this system frequently" whereas statement #2 is "I found this system unnecessarily complex". The participant's scores for each question are converted to a new number, added together, and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  SUS scores above 68 are considered above average and anything below 68 is below average.
Trail Making Test - Digital | Change from baseline at 3 months
  This is a standardized test of cognitive function. The test consists of two Trails, Trail A and Trail B. Trail A requires the participant to tap on 25 numbers on the screen in order from smallest to largest (1, 2, 3, etc). Trail B requires participants to tap on alternative numbers and letters in consecutive order from smallest/first to largest/last (1, A, 2, B, 3, C etc).
Trail Making Test - Digital | Change from baseline at 6 months
  This is a standardized test of cognitive function. The test consists of two Trails, Trail A and Trail B. Trail A requires the participant to tap on 25 numbers on the screen in order from smallest to largest (1, 2, 3, etc). Trail B requires participants to tap on alternative numbers and letters in consecutive order from smallest/first to largest/last (1, A, 2, B, 3, C etc).
Trail Making Test - Digital | Change from baseline at 9 months
  This is a standardized test of cognitive function. The test consists of two Trails, Trail A and Trail B. Trail A requires the participant to tap on 25 numbers on the screen in order from smallest to largest (1, 2, 3, etc). Trail B requires participants to tap on alternative numbers and letters in consecutive order from smallest/first to largest/last (1, A, 2, B, 3, C etc).
Trail Making Test - Digital | Change from baseline at 12 months
  This is a standardized test of cognitive function. The test consists of two Trails, Trail A and Trail B. Trail A requires the participant to tap on 25 numbers on the screen in order from smallest to largest (1, 2, 3, etc). Trail B requires participants to tap on alternative numbers and letters in consecutive order from smallest/first to largest/last (1, A, 2, B, 3, C etc).
Modified Fear of Falling Avoidance Behavior Questionnaire | Change from baseline at 3 months
  This is a standardized self-report assessment that measures behaviors that may be avoided due to a fear of falling
Modified Fear of Falling Avoidance Behavior Questionnaire | Change from baseline at 6 months
  This is a standardized self-report assessment that measures behaviors that may be avoided due to a fear of falling
Modified Fear of Falling Avoidance Behavior Questionnaire | Change from baseline at 9 months
  This is a standardized self-report assessment that measures behaviors that may be avoided due to a fear of falling
Modified Fear of Falling Avoidance Behavior Questionnaire | Change from baseline at 12 months
  This is a standardized self-report assessment that measures behaviors that may be avoided due to a fear of falling
Depression Screen | Change from baseline at 3 months
  The Depression Screen is a 2-item questionnaire that asks about how the person has been feeling over the past 2 weeks.
Depression Screen | Change from baseline at 6 months
  The Depression Screen is a 2-item questionnaire that asks about how the person has been feeling over the past 2 weeks.
Depression Screen | Change from baseline at 9 months
  The Depression Screen is a 2-item questionnaire that asks about how the person has been feeling over the past 2 weeks.
Depression Screen | Change from baseline at 12 months
  The Depression Screen is a 2-item questionnaire that asks about how the person has been feeling over the past 2 weeks.
Adherence to Exercise Program (Intervention Group Only) | through study completion, an average of 1 year
  Average number of days per week the exercise program was completed
Total number of repetitions of all exercises completed | through study completion, an average of 1 year
  Total number of repetitions of all exercises completed
Adherence to Education Modules | through study completion, an average of 1 year
  Total number of education modules completed

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, PhD, Study Director — Texas A&M University
Locations (1):
- Blue Marble Health, Altadena, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared